CLINICAL TRIAL: NCT03369262
Title: A Phase 2a, Double-blind, Parallel Group, Randomised, Placebo Controlled, Proof of Concept Study to Assess the Efficacy, Safety and Pharmacokinetics of OBE022 added-on to Atosiban, After Oral Administration in Pregnant Women With Threatened Spontaneous Preterm Labour
Brief Title: PoC Study of OBE022 in Threatened Preterm Labour
Acronym: PROLONG
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: ObsEva SA (Industry)
Collaborators: Scope International AG (Industry); Iqvia Pty Ltd (Industry); Cytel Inc. (Industry); PhinC Development (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 17-OBE022-003
Record Dates: First submitted 2017-11-30; First posted 2017-12-11 (Actual); Last update posted 2021-06-07 (Actual); Status verified 2021-06

CONDITIONS: Preterm Labor
Keywords: preterm labor; preterm birth; premature birth; tocolysis; prostaglandin F2α antagonist; PGF2α; tocolytic
MeSH Terms: conditions — Obstetric Labor, Premature; Premature Birth | interventions — obe022; atosiban

STUDY DESIGN:
Intervention Model Description: A phase 2a, double-blind, parallel group, randomised, placebo controlled, added-on to atosiban.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Matching placebo.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active (Experimental): OBE022 plus atosiban:
  OBE022 will be given orally from Day 1 to Day 7. OBE022 treatment will be initiated ideally simultaneously or at a maximum within 24 h after atosiban start.
  * Loading dose: 1 000 mg on Day 1.
  * Maintenance dose on Day 1: 500 mg in the evening if loading dose was administered in the morning. If loading dose was administered in the afternoon, then the next dose will take place on the morning of Day 2.
  * Maintenance dose from Day 2 to Day 7: 500 mg twice a day (only morning dose on Day 7)
  Atosiban will be administered over 48h as per label.
  Interventions: Drug: OBE022; Drug: Atosiban
- Placebo (Active Comparator): OBE022 matching placebo plus atosiban:
  OBE022 matching placebo administration will follow the same regimen as the active group.
  Atosiban will be administered over 48h as per label.
  Interventions: Drug: Placebos; Drug: Atosiban

INTERVENTIONS:
Drug: OBE022 — Oral
  Arms: Active
Drug: Placebos — Oral
  Arms: Placebo
Drug: Atosiban — I.V.

SUMMARY:
This is a proof-of-concept study in 2 parts.

In Part A, patients will receive OBE022 open-label in order to assess the safety and pharmacokinetics in pregnant women with spontaneous preterm labour with a gestational age between 28 0/7 and 33 6/7 weeks.

Part B has a double-blind, randomised, placebo controlled, parallel group and multicentre design and will assess the efficacy, safety and pharmacokinetics in pregnant women with threatened spontaneous preterm labour with a gestational age between 24 0/7 and 33 6/7 weeks.

All patients in part A and part B must receive atosiban infusion for 48 hours as standard of care treatment. Patients from Part A will receive OBE022 open label. Patients from Part B will be randomised to receive OBE022 or matching placebo. IMP treatment duration will be up to 7 days. IMP treatment will be stopped in case of delivery prior to Day 7.

ELIGIBILITY:
Key Inclusion Criteria:

Part A

* Pregnant females aged ≥ 18 years
* Patients with a singleton or twin pregnancy
* Gestational age between 28 0/7 and 33 6/7
* Administered or prescribed atosiban for the treatment of preterm labour

Part B

* Pregnant females aged ≥ 18 years
* Patients with a singleton or twin pregnancy
* Gestational age between 24 0/7 and 33 6/7
* Administered or prescribed atosiban for the treatment of preterm labour
* ≥4 uterine contractions per 30 minutes
* Cervical dilatation of 1 to 4 cm inclusive
* At least one of the following signs of preterm labour:

  1. positive IGFBP-1 or fœtal Fibronectin test
  2. cervical length ≤ 25mm
  3. progressive cervical change

Key Exclusion Criteria:

* Fœtal death in utero in current or previous pregnancy after gestational week 24 or expected high risk of fœtal death in the coming days
* Oligohydramnios
* Known pathological Doppler ultrasound of the umbilical artery
* Any contraindications for the mother or the fœtus to stop labour or prolong pregnancy or any maternal or fœtal conditions likely to indicate iatrogenic delivery in the next 7 days, including but not limited to:

  1. Premature rupture of membranes
  2. Evidence or suspicion of abruptio placenta
  3. Signs and/or symptoms of chorio-amnionitis
  4. Pre-eclampsia, eclampsia or HELLP-syndrome
* Use of cervical cerclage in the current pregnancy or a pessary in situ
* Current use of anti-hypertensive medication
* Treatment with other tocolytics within specified time before the baseline assessment of uterine contractions

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2018-01-10 (Actual); Primary Completion 2020-07-08 (Actual); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Incidence of delivery within 2 days (48 h) from start of IMP administration | 48 hours
Incidence of delivery within 7 days (168 h) from start of IMP administration | 168 hours
Incidence of delivery before 37 weeks of GA | Up to 13 weeks from start of IMP administration
Time to delivery measured from start of IMP administration | Up to 17 weeks from start of IMP administration

OTHER OUTCOMES:
Maternal incidence of AEs from Day 1 until 28 days after birth. | 28 days after birth
Maternal incidence of TEAEs from Day 1 until 28 days after birth. | 28 days after birth
Maternal incidence of clinically significant changes in laboratory safety tests, from Day 1 until 28 days after birth. | 28 days after birth
Maternal incidence of clinically significant changes in vital signs, from Day 1 until 28 days after birth. | 28 days after birth
Incidence of AEs indicating fœtal distress such as growth retardation and/or changes in fœtal heart rate monitoring and/or amniotic fluid index (AFI) from Day 1 to Day 7 and Day 14 (or earlier if birth). | Up to 14 days after start of IMP administration
In Part A only: Incidence of fœtal adverse events in relation with the cardiovascular function assessed by Doppler ultrasound on Day 1 to 3 and Day 7 from IMP start. | Up to 7 days after start of IMP administration
Incidence of infants experiencing adverse events from birth until 28 days after birth. | Up to 28 days after birth
Incidence of infants experiencing clinical significant changes in vital signs from birth until 28 days after birth. | Up to 28 days after birth
Apgar score. | At birth, at 1 minute and 5 minute
  The score is a rapid method for assessing a neonate immediately after birth. Elements of the Apgar score include color, heart rate, reflexes, muscle tone, and respiration, each weighted evenly and assigned a value of 0, 1, or 2. The components are then added together to give a total score (0 to 10) that is recorded at 1 and 5 minutes after birth.
Weight. | At birth and 28 days after birth.
Head circumference. | At birth and 28 days after birth.
Incidence of infants experiencing prematurity-related events | At birth.
Incidence of duration of hospitalization and or re-admission to hospital. | Up to 28 days after birth.
Incidence of infants with one or more Ages and Stages Questionnaire® domain score(s) below the cut-off score at 6 months, 12 months and 24 months of age, adjusted for gestational age at birth. | Up to 24 months
  The Ages and Stages Questionnaire (ASQ) is a parent-completed questionnaire designed to be used as a general developmental screening tool. The ASQ-3 covers five areas of child development that includes: personal social, gross motor, fine motor, problem solving, and communication. Parents complete the questionnaire independent of professionals, indicating for each item "yes" if child performs the item, "sometimes" indicating an occasional or emerging skill, or "not yet" indicating that the child does not yet perform the behavior
Plasma concentration of OBE022/OBE002 at Day 1, Day 2, Day 3 and Day 7. | Up to 7 days after start of IMP administration
Pharmacokinetic parameters of OBE022/OBE002 at Day 7 | Day 7
  Area under the curve (AUC)
Pharmacokinetic parameters of OBE022/OBE002 at Day 7 | Day 7
  Maximal concentration (Cmax)
Pharmacokinetic parameters of OBE022/OBE002 at Day 7 | Day 7
  Half-life.
Fœtal (cord blood)-maternal OBE002 concentration ratio at the time of delivery for patients who received IMP treatment within the previous 24 h. | Day of delivery
Changes in uterine contractions as assessed by electrohysterography, tocodynamometry or abdominal palpation at each hour during the first 6 hours after IMP start. | Up to 6 hours after IMP start.

CONTACTS AND LOCATIONS:
Locations (18):
- Czechia (3):
  - Gynekologicko-porodnická klinika Fakultní nemocnice Brno, Brno
  - Gynekologicko-porodnická klinika 1. LF UK a VFN v Praze, Prague
  - Ústav pro péči o matku a dítě, Prague
- Helsinki Universisty Hospital, Helsinki, Finland
- Israel (4):
  - Hilel Yafe Medical Center, Maternal Fetal Unit, Haifa
  - Rambam Medical Center, Maternal Fetal Unit, Haifa
  - Meir Medical Center, Obstetrics and Gynecology Department, Kfar Saba
  - Rabin Medical Center, Fetal-Maternal Medicine, Helen Schneider's Hospital for Women, Petah Tikva
- Russia (4):
  - Moscow Regional Perinatal Center, Balashikha
  - Kazan State Medical University, Kazan'
  - City clinical hospital № 15 named after O. M. Filatov of Healthcare Department of Moscow, Moscow
  - Perinatal center of the City Clinical Hospital #24, Moscow
- Spain (4):
  - Hospital La Paz, Madrid
  - Hospital Clínico Universitario Virgen de la Arrixaca, Murcia
  - Hospital Clínico Universitario de Santiago, Santiago de Compostela
  - Hospital Universitari i Politècnic La Fe, Valencia
- Vietnam (2):
  - Hanoi Obstetrics and Gynecology Hospital, Hanoi
  - My Duc Hospital, Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wilson A, Hodgetts-Morton VA, Marson EJ, Markland AD, Larkai E, Papadopoulou A, Coomarasamy A, Tobias A, Chou D, Oladapo OT, Price MJ, Morris K, Gallos ID. Tocolytics for delaying preterm birth: a network meta-analysis (0924). Cochrane Database Syst Rev. 2022 Aug 10;8(8):CD014978. doi: 10.1002/14651858.CD014978.pub2. PMID 35947046